CLINICAL TRIAL: NCT00574561
Title: Magnetocardiography (MCG) in Subjects Undergoing CT Angiography (CTA)
Status: Withdrawn | Type: Observational
Why Stopped: sponsor funding
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: CardioMag Imaging (Industry)
Responsible Party: Kirsten Tolstrup, MD, Cedars-Sinai Medical Center
Other Study IDs: 10057
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Chest Pain
Keywords: CT angiography (CTA); Magnetocardiography (MCG); heart disease
MeSH Terms: conditions — Chest Pain; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators wish to study the magnetic field map using magnetocardiography (MCG) in subjects undergoing computed tomographic angiography (visualization of the heart arteries using CT scanning, CTA). The main purposes is to investigate if MCG is capable of detecting the presence of obstructive coronary artery disease (CAD) as detected by CT angiography (CTA) as well if the MCG can exclude the presence of CAD as defined by CTA.

Secondarily the investigators will look at the correlation of MCG with non-obstructive CAD and the correlation of MCG with other tests (treadmill testing, stress echo or nuclear scan, coronary angiography) done as part of the work up for CAD.

DETAILED DESCRIPTION:
Cardiomagnetism refers to the detection, analysis and interpretation of the magnetic fields generated by the electrical activity of the heart. The peak value of the magnetic fields of the heart is more than a million times smaller than the Earth's magnetic field. A major breakthrough in the capability of measuring such small fields came with the invention of the SQUID (superconducting quantum interference device) in the late sixties. The first magnetocardiograms (MCGs) measured with the SQUID were recorded by Cohen et al. in 1970. These earlier measurements were performed in very expensive magnetically shielded rooms, initially utilizing only one or two SQUID probes. In the eighties this technology was tested in several laboratories creating a magnetic field map by moving one SQUID sequentially above the chest to create an image of the whole hearts magnetic field. These maps were then attempted correlated with various pathologies (1).

Since then the technology has been greatly improved and several multi-channel machines are in use across the world for research purpose for arrhythmia localization and ischemia detection. However, at present time, only one company (CardioMag Imaging, Schenectady, New York) has developed a machine that operates outside a shielded room.

The CardiomagImaging (CMI) Magnetocardiograph (MCG) is capable of noninvasive recording of magnetic fields arising from the electrical activity of the heart with very high spatial and temporal resolution. The temporal trace of the MCG is analogous to an ECG, and, similarly, can be recorded in multiple leads. This MCG device has been specifically developed for the general purpose (outside shielded room) of non-contact, non-invasive diagnostics of ischemia.

The CMI MCG device has been approved by the FDA as a safe tool to measure and record the magnetic field arising from the heart's electrical currents. It is awaiting FDA approval for the specific diagnosis of ischemia in chest pain patients (2,3).

We have been using the CMI 9-channel MCG for detection of ischemia in patients admitted to Cedars-Sinai Medical Center for acute chest pain syndrome. The results are very exciting and have been published in abstracts and one manuscript, with another manuscript in submission (4,5). In summary, we studied 75 patients with acute chest pain and 65 healthy volunteers and found a very strong association with an abnormal MCG scan and ischemia (p<0.0001). The sensitivity, specificity, PPV and NPV was 87.1%, 85.7%, 64.3%, and 95.7%, respectively. In comparison, the diagnostic value of the stress SPECT imaging was 91.3%, 75.0%, 75.0%, and 91.3%, for sensitivity, specificity, positive and negative predictive value, respectively. These results were achieved without the use of stress provocation, contrast administration, or any ionizing radiation, and the results were available immediately.

Since starting the chest pain protocol another diagnostic imaging technology has become more widespread used, 64-slice CT angiography. This technology utilizes a fast CT scanner and involves administration of a contrast agent, but avoids the invasiveness of a heart catheterization. The accuracy of detection of CAD and its exclusion is very high as compared with angiography (6). Although minimally invasive, the CT angiogram does involve a radiation dose similar to that used with stress nuclear testing, approximately 900 to 1100 mrem (6) and the iodine contrast used may cause contrast nephropathy, especially in diabetics and those with already impaired renal function. The use of this technology provides an opportunity to find subjects with normal coronary arteries with accuracy close to as high as for invasive coronary angiography. To date, this population has been hard to study, since subjects with a normal stress test rarely will undergo more invasive studies.

Therefore, we wish to conduct this correlative study with CT angiography and the entirely noninvasive and risk free MCG to see if we in the future may be able to avoid some of the risks associated with CTA. We think that we may find that subjects with a clearly abnormal MCG may not need CTA, but could proceed directly to angiography and possible angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing 64-slice CT angiography

Exclusion Criteria:

* Hemodynamically unstable patients
* Patients with pacemakers or internal defibrillators
* Minors < 18 years of age
* Patients unable to lie flat for the examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing CT angiography to evaluate their coronary arteries for the presece of heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Tolstrup, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] 1)Stroink G, MacAuley C, Montague TJ, Horacek BM. Normal and abnormal components in magnetocardiographic maps of a subject with myocardial infarction. Med. Biol. Eng. Comp. 1985, 23, 61-62.
- [Background] Koch H. Recent advances in magnetocardiography. J Electrocardiol. 2004;37 Suppl:117-22. doi: 10.1016/j.jelectrocard.2004.08.035. PMID 15534820
- [Background] Fenici R, Brisinda D, Meloni AM. Clinical application of magnetocardiography. Expert Rev Mol Diagn. 2005 May;5(3):291-313. doi: 10.1586/14737159.5.3.291. PMID 15934809
- [Background] 4)Tolstrup K, Madsen B, et al. Resting Magnetocardiography Accurately Detects Myocardial Ischemia in Chest Pain Patients with normal or non-specific ECG Findings. Cardiology. 2006;106:270-276.
- [Background] 5)Kirsten Tolstrup, Donatella Brisinda, Anna M. Meloni, Brian Cheung, Sean Rashti, Robert J. Siegel, Riccardo Fenici. Resting Magnetocardiography is Highly Accurate for the Detection of Ischemia in Patients with Acute Chest Pain Syndrome. Submitted.
- [Background] Stein PD, Beemath A, Kayali F, Skaf E, Sanchez J, Olson RE. Multidetector computed tomography for the diagnosis of coronary artery disease: a systematic review. Am J Med. 2006 Mar;119(3):203-16. doi: 10.1016/j.amjmed.2005.06.071. PMID 16490463